CLINICAL TRIAL: NCT03132311
Title: Immunogenicity and Safety of the Yellow Fever Vaccine in HIV Infected Individuals
Acronym: YF-HIV
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections
Keywords: yellow fever vaccine; hiv
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV positive subjects (Experimental): 300 HIV positive adults with CD4 > 200 cells/mm3, stratified in 3 groups (100 patients in each group) according to CD4 counts (200-350; 351-500, >500 cells/mm3).
  Assigned intervention: Yellow fever vaccination (17 DD Biomanguinhos)
  Interventions: Biological: Yellow Fever vaccination (17 DD Biomanguinhos)
- HIV negative subjects (Active Comparator): 100 HIV negative adults.
  Assigned intervention: Yellow fever vaccination (17 DD Biomanguinhos)
  Interventions: Biological: Yellow Fever vaccination (17 DD Biomanguinhos)

INTERVENTIONS:
Biological: Yellow Fever vaccination (17 DD Biomanguinhos) — One intramuscular injection

SUMMARY:
Phase 4 study to evaluate the immunogenicity and Safety of the 17DD Yellow Fever vaccine in HIV infected individuals, compared to non-HIV-infected individuals.

Main objective:

To compare the proportion of seroconversion and the geometric mean of neutralizing antibodies 30 days and 365 days after vaccine.

Secondary objectives:

To evaluate whether the titles of neutralizing antibodies are associated with CD4 lymphocyte counts, CD8 lymphocyte counts, CD4 nadir, HIV viral load and use of antiretroviral therapy. To assess the yellow fever vaccine viremia at day 10 after vaccine.To compare the incidence of adverse events in HIV-infected and non-HIV-infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected adults, age >= 18 and <60 years old.
* CD4 > 200 cells/mm³ within the last 6 months prior to inclusion. Individuals with no CD4 results in the last 6 months which have undetectable HIV viral load and last CD4 count > 350 can be included.
* Healthy HIV-uninfected individuals (aged >= 18 and < 60)
* No history of Yellow Fever vaccination
* Willing to participate and to sign the consent

Exclusion Criteria:

* Individuals with chronic diseases such as: decompensated diabetes, kidney failure (in dialysis), liver failure/cirrhosis, cancer (except for non-melanoma skin cancer and in situ HIV related carcinoma), use of immunosuppressive agents (including prednisone ≥ 20mg/day, during 7 or more days in the last 30 days before inclusion).
* Pregnant women
* Hypersensitivity reaction to eggs, chicken protein. Allergy to erythomycin or kanamycin. Hereditary fructose intolerance.
* Administration of immunoglobulins or blood derivates < 3 months or life attenuated vaccine <1 month.
* History of thymic dysfunction (including thymoma and thymectomy).
* Use of anti-CCR5
* symptoms of severe acute illnesses or fever (axillary temperature ≥ 38°C)
* HIV positive rapid test for HIV negative subjects.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity | 30 days after the vaccine
  Seroconversion
Immunogenicity | 30 days after the vaccine
  Neutralizing antibodies titers
Immunogenicity | 365 days after the vaccine
  Seroconversion
Immunogenicity | 365 days after the vaccine
  Neutralizing antibodies titers

SECONDARY OUTCOMES:
Viremia | 7 days after the vaccine
  Yellow Fever vaccine viremia
Adverse events | up to 30 days after the vaccine
  Yellow Fever vaccine related adverse events
Immunogenicity | 5 years after the vaccine
  Neutralizing antibodies titles
Immunogenicity | 10 years after the vaccine
  Neutralizing antibodies titles

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macieira KV, Caetano DG, De Lima SMB, Wagner Giacoia-Gripp CB, Cortes FH, Da Silva Cazote A, De Souza Azevedo Soares A, Dos Santos Alves N, De Souza Borges Quintana M, Costa M, Brandao LGP, De Andrade MM, Grinsztejn B, Coelho LE, De Almeida DV. Differential gene expression of cytokines, receptors, and miRNAs in individuals living with HIV-1 and vaccinated against yellow fever. Mol Immunol. 2023 Dec;164:58-65. doi: 10.1016/j.molimm.2023.10.013. Epub 2023 Nov 10. PMID 37952362
- [Derived] Motta E, Camacho LAB, Cunha M, de Filippis AMB, Lima SMB, Costa M, Pedro L, Cardoso SW, Cortes FH, Giacoia-Gripp CBW, Morata M, Nazer S, Moreira RI, de Oliveira Souza MC, Mendes YS, Souza Azevedo A, Dos Santos Alvez N, Grinsztejn B, Coelho LE. Immunogenicity and reactogenicity of yellow fever vaccine in people with HIV. AIDS. 2023 Dec 1;37(15):2319-2329. doi: 10.1097/QAD.0000000000003696. Epub 2023 Aug 23. PMID 37650759